CLINICAL TRIAL: NCT07031206
Title: Investigating Pre-Procedural Anxiety and Effect of Analgesia on Intrauterine Device Placement and Endometrial Biopsy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pamela Berens, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-25-0136
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Pain
Keywords: intrauterine device (IUD) insertion; endometrial biopsy (EMB)
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Epinephrine; Hydroxyzine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Paracervical block- Lidocaine without epinephrine with Hydroxyzine hydrochloride if needed (Experimental)
  Interventions: Drug: Paracervical block- Lidocaine without epinephrine; Drug: Hydroxyzine Hydrochloride
- Benzocaine Gel applied to the cervix with Hydroxyzine hydrochloride if needed (Experimental)
  Interventions: Drug: Benzocaine Gel applied to the cervix; Drug: Hydroxyzine Hydrochloride
- No analgesia with Hydroxyzine hydrochloride if needed (Experimental)
  Interventions: Drug: Hydroxyzine Hydrochloride

INTERVENTIONS:
Drug: Paracervical block- Lidocaine without epinephrine — 1-2 cc of Lidocaine at the tenaculum site on the cervix at 12 o-clock will be injected after pain scale #1 is completed. Pain scale #2 will be done then 3 cc of 1% lidocaine at 4 and 8 o'clock position of the cervix will be administered. The IUD insertion or EMB will be performed nd pain scale #3 will be done.
  Arms: Paracervical block- Lidocaine without epinephrine with Hydroxyzine hydrochloride if needed
Drug: Benzocaine Gel applied to the cervix — After pain scale #1 is performed , topical benzocaine will be applied to the cervix with Procto swabs and this will be allowed to remain on cervix for 203 minutes. Then Betadine will be applied to the cervix and surrounding vaginal tissue followed by pain scale #2. IUD insertion or EMB will be done followed by pain scale #3.
  Arms: Benzocaine Gel applied to the cervix with Hydroxyzine hydrochloride if needed
Drug: Hydroxyzine Hydrochloride — Preprocedure, a GAD 7 scoring will be performed to determine level of anxiety. If > 10 indicating Moderate anxiety, participants will be offered pretreatment with Anxiolytic (Hydroxyzine 25mg) approximately 15-20 mins before procedure. If this is done at the preceding visit, participants will be sent home with a prescription for hydroxyzine to be taken 10-15 mins before the procedure when participants are brought back for procedure visit.

SUMMARY:
The purpose of this study is to evaluate pre-procedural anxiety and patient pain perception with IUD insertion/ EMB procedure when using analgesia versus no analgesia by the end of the study and to evaluate the effect of age, race, parity, type of IUD and anxiety on pain and to offer better pain management in our patient population, undergoing IUD insertion/EMB procedure at the end of our study.

ELIGIBILITY:
Inclusion Criteria:

* present for an IUD insertion procedure and/or for EMB procedure.

Exclusion Criteria:

* current Pelvic inflammatory disease (PID)
* contraindications to IUD or EMB
* malignancy
* contraindication to hydroxyzine/Lidocaine/Benzocaine
* positive pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in pain perception during IUD insertion as assessed by the Faces Pain Visual Analogue Scale (VAS) | baseline (with the speculum in place before pain management procedures), after tenaculum placement (but before IUD placement or EMB) and immediately after IUD insertion or EMB.
  VAS is scored from 1-10, higher score indicating greater pain

SECONDARY OUTCOMES:
Change in anxiety as assessed by the General Anxiety Disorder-7 (GAD-7) scale | baseline, and after taking Hydroxyzine about 15-30 mins before procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Berens, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No